CLINICAL TRIAL: NCT04386018
Title: A Registered Cohort Study on Natural Course and Drug Efficacy of Inflammatory Demyelination Disease
Brief Title: A Registered Cohort Study of Inflammatory Demyelination Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ning Wang, MD., PhD. (Other)
Responsible Party: Sponsor-Investigator, Ning Wang, MD., PhD., Director, First Affiliated Hospital of Fujian Medical University
Organization: First Affiliated Hospital of Fujian Medical University (Other)
Other Study IDs: MRCTA,ECFAH of FMU [2019]216
Record Dates: First submitted 2020-05-10; First posted 2020-05-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Demyelinating Autoimmune Diseases, CNS
MeSH Terms: conditions — Demyelinating Autoimmune Diseases, CNS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will provide further insights into the natural course of Inflammatory demyelination disease including clinical features，progression, related antibody spectrum and drug treatment effect

ELIGIBILITY:
Inclusion Criteria:

1. Outpatient or inpatient
2. Meet the diagnostic criteria of Inflammatory Demyelination Disease.
3. Voluntary participation and informed consent signed by the applicant or his/her family.

Exclusion Criteria:

1. Severe complications
2. Poor prognosis (<1 year survival)
3. Severe mental disorder and inability to cooperate with the examination.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Inflammatory Demyelination Disease who are diagnosied in the First Affiliated Hospital of Fujian Medical Universtiy by two neurolgists
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-05-15 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
The correlation between clinical phenotypes and Serum antibodies | from date of enrollment until the date of death from any cause,assessed up to 20 years
  Different clinical subtypes of Demyelinating Autoimmune Diseases have different course and prognosis.It may be related to different serum antibodies.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology,First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China